CLINICAL TRIAL: NCT03968783
Title: The Effect of Suturing Material on Scar Healing; a Randomised Controlled Trial
Brief Title: The Effect of Suturing Material on Scar Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Cesarean suture study
Record Dates: First submitted 2019-05-28; First posted 2019-05-30 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Wound Heal; Cesarean Section Complications; Cesarean Wound Disruption; Suture Related Complication
Keywords: cesarean section; scar heal; isthmocele; suture material; saline infusion sonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monofilament suture (Experimental): continuous double-layer unlocked suturing with 1.0 monofilament synthetic absorbable suture
  Interventions: Other: Monofilament suture
- Multifilament suture (Active Comparator): continuous double-layer unlocked suturing with 1.0 multifilament synthetic absorbable suture
  Interventions: Other: Multifilament suture

INTERVENTIONS:
Other: Monofilament suture — 1.0 monofilament synthetic absorbable suture for closure of the low transverse uterine incision
  Arms: Monofilament suture
Other: Multifilament suture — 1.0 multifilament synthetic absorbable suture for closure of the low transverse uterine incision
  Arms: Multifilament suture

SUMMARY:
We want to compare the effects of 2 suture materials (monofilament and multifilament) on healing of the uterine scar after a cesarean delivery.

DETAILED DESCRIPTION:
Cesarean section (CS) is the most common type of obstetric surgery. When medically justified, CS can effectively prevent maternal and perinatal mortality and morbidity however, there are many short and long-term complications of CS. One of the most common complications is the CS scar defect. CS scar defects can develop after transverse incision of the lower uterine segment, which may result in prolonged postmenstrual bleeding, spotting, pelvic pain, and infertility. Suture material is an essential part of any major surgery, serving to hold opposing tissues together and accelerate the healing process, resulting in decreased scarring of the affected areas. We sought to evaluate the effects of different synthetic absorbable suture materials on cesarean scar defect formation.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy at term >37 weeks of gestational age

Exclusion Criteria:

* history of previous cesarean section
* history of previous uterine surgery
* multiple gestation, placenta previa, polyhydramnious, fetal macrosomia
* uterine atony history
* gestational diabetes mellitus, gestational hypertension, preeclampsia, current or previous history of heart disease, liver, renal disorders or known coagulopath
* active labor (with regular uterine contractions and cervical dilatation >4 cm

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 95 (Actual)
Dates: Start 2019-05-27 (Actual); Primary Completion 2019-07-27 (Actual); Study Completion 2020-01-27 (Actual)

PRIMARY OUTCOMES:
The healing ratio | 6 months
  Six months after the operation, the integrity of the cesarean scar at the uterine incision site will be assessed by hydrosonography. The healing ratio will be calculated as the thickness of the residual myometrium covering the defect, divided by the sum of the thickness of the residual myometrium covering the defect and the height of the wedge-shaped defect.

SECONDARY OUTCOMES:
blood loss | 24 hours
  The hemoglobin and hematocrit values will be measured 24 hours after CS
additional sutures | 2 hours
  number of additional hemostatic sutures

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakıf University Hospital, Istanbul, Turkey (Türkiye)